CLINICAL TRIAL: NCT04164329
Title: Anesthetic Neurotoxicity: the Association Between General Anesthesia and the Level of Plasma Neurofilament Light
Acronym: ANESTOX-2019
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiocentro Ticino (Other)
Responsible Party: Principal Investigator, Tiziano Cassina, Professor med. Tiziano Cassina, Cardiocentro Ticino
Other Study IDs: 2019-01739
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: General Anesthetics Toxicity
Keywords: Neurotoxicity; anesthesia; Neurofilament Light
MeSH Terms: conditions — Neurotoxicity Syndromes; Charcot-Marie-Tooth disease, Type 1F | interventions — Anesthetics, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: The exposed group will be composed by the patients that undergo CRT/ICD implantation (general anesthesia).
  Interventions: Drug: General anesthetic
- Not exposed group: The non-exposed group, or control group, will be composed by the patients undergo PM implantation (without anesthesia)

INTERVENTIONS:
Drug: General anesthetic — General anesthesia (propofol, fentanyl, sevorane, remifentanyl, rocuronium)
  Groups: Exposed group

SUMMARY:
A prospective controlled single centre study designed to determine the association between the exposure to anesthetic agents and the pre and postoperative changes in plasma Neurofilament Light levels, biomarkers of neurological injury, in patients with similar surgical intervention but different anesthetic techniques.

Secondary endpoints: Association between the changes in plasma Neurofilament Light levels and the development of post-operative neurocognitive disorders as acute delirium.

DETAILED DESCRIPTION:
Our intent is to evaluate the impact of the general anesthesia on the Central Nervous System, trying to minimize the surgical bias as much as possible. For this purpose, it is necessary to consider two groups of patients who undergo to similar surgical intervention, but with exposed to different anesthetic techniques. In particular, one group with local anesthesia and one group with general anesthesia.

The population sample will be composed of all patients who satisfy the inclusion and exclusion criteria and scheduled for the implantation of pacemaker (PM) - a procedure that require a local anesthesia - and the implantation of a cardioverter defibrillator (ICD), a cardiac resynchronization therapy pacemaker (CRT-P) and a cardiac resynchronization therapy defibrillator (CRT-D) at the Cardiocentro Ticino Lugano, procedures usually realize under general anesthesia.

The population sample will be divided in two groups: the non-exposed group, or control group, will be composed by the patients undergo PM implantation (without anesthesia) and the exposed group will be composed by the patients that undergo CRT/ICD implantation (general anesthesia).

Inclusion criteria:

* Same type of surgery: ICD,CRT-P, CRT-D and PM implantation;
* Age > 18 years old
* Patients who have expressed their consent to the participation of the study

Exclusion criteria:

- Patients with history of neurodegenerative diseases and neurocognitive disorders: the presence of these disorders could influence the level of the neuro-markers.

No change will be applied to normal clinical practice: we'll collect two blood samples, taken from routine samples already performed in our clinical practice, for the dosage of Neurofilament Light plasma levels before (t0) and after the procedure (t+24h).

Our intent is to compare the NF-L plasma levels delta (pre or t0 - postoperative or t24) between the exposed group (general anesthesia) and the not exposed group (local anesthesia).

Blood samples will be collected and stored in EDTA at the times specified above and anonymized. The samples, post anonymization, will be send to the University Hospital of Basel (Basel, Switzerland) where the plasma concentration of neurodegeneration markers will be blindly measured using the SiMoA neurology 4-plex assay.

The neurological status of the patients will be monitored daily during the first 2 days of the post-operative course in intensive care or in the ward. The screening of the phenomenon will be carried out by the nursing staff through the CAM-ICU and CAM (screening), in accordance with the internal protocols. The screening will be performed and documented at least three times a day or when the need is detected by the nursing staff. Any diagnosis of delirium will be certified by the neurologist.

Exams or procedures that differ from normal clinical practice will not be performed, except for the dosage of Neurofilament Light.

ELIGIBILITY:
Inclusion Criteria:

* Same type of surgery: ICD,CRT-P, CRT-D and PM implantation;
* Age > 18 years old
* Patients who have expressed their consent to the participation of the study

Exclusion Criteria:

- Patients with history of neurodegenerative diseases and neurocognitive disorders: the presence of these disorders could influence the level of the neuro-markers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population sample will be composed of all patients who satisfy the inclusion and exclusion criteria and scheduled for the implantation of pacemaker (PM) - a procedure that require a local anesthesia - and the implantation of a cardioverter defibrillator (ICD), a cardiac resynchronization therapy pacemaker (CRT-P) and a cardiac resynchronization therapy defibrillator (CRT-D) at the Cardiocentro Ticino Lugano, procedures usually realize under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma Neurofilament Light levels | 24 hours
  Comparison of changes in plasma Neurofilament Light levels pre and postoperative in patients exposed and not exposed to general anesthesia.

SECONDARY OUTCOMES:
Changes in plasma Neurofilament Light levels and acute postoperative neurocognitive disorders | 48 hours
  Association between the changes in plasma Neurofilament Light levels and the development of post-operative neurocognitive disorders as acute delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Tiziano TC Cassina, Professor, Principal Investigator — Cardiocentro Ticino; Stefania SB Buson, Dr.ssa, Principal Investigator — Cardiocentro Ticino
Locations (1):
- Cardiocentro Ticino, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No